CLINICAL TRIAL: NCT05261308
Title: New Polyamide Prosthesis for Treatment of Non-union Mid Shaft Clavicle Fracture: A Case Report
Brief Title: Customized Polyamide Prosthesis. for Mid Shaft Clavicle Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sahar Ahmed Abdalbary, Associate professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: polyamide
Record Dates: First submitted 2022-02-04; First posted 2022-03-02 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Treatment Adherence and Compliance
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- prosthesis (Experimental): The polyamide prosthesis
  Interventions: Other: new prosthesis

INTERVENTIONS:
Other: new prosthesis — Operation to fix the new prosthesis

SUMMARY:
Herein we describe the management of a patient who presented with progressive brachial plexopathy following the initial nonoperative management of a mid shaft clavicular fracture by using 3 D customized polyamide prosthesis.

DETAILED DESCRIPTION:
we made surgery to fix the new polyamide prosthesies in the clavicle.

ELIGIBILITY:
Inclusion Criteria:

* fracture midshaft clavicle

Exclusion Criteria:

* normal clavicle

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
American shoulder and elbow surgeons score Special Score for shoulder pain and function | after 2 and half years
  American shoulder and elbow surgeons score Special Score for shoulder pain and function.
  The American shoulder and elbow surgeons score is a composite instrument, requiring both a physician assessment and a patient-completed portion.
  . This includes a section on pain (7 items) and a section on activities of daily living (10 items). Scores range from 0 to 100 with a score of 0 indicating a worse shoulder condition and 100 indicating a better shoulder condition.
  Intensity of pain: 0; Putting on a coat is not difficult; Sleeping on the affected side is not difficult; Washing my back/doing up my bra is not difficult; Managing toiletting is not difficult; Combing my hair is not difficult; Reaching a high shelf is not difficult; Lifting 10lbs. (4.5kg) above my shoulder is not difficult; Throwing a ball overhand is not difficult; Doing my usual work is not difficult; Doing my usual sport/leisure activity is not difficult; It means good shoulder

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Abdalbary, professor, Principal Investigator — Nahda University, Faculty of Physical Therapy
Locations (2):
- Egypt (2):
  - Sahar Abdalbary, Cairo, Select State/province
  - Sahar, Cairo

IPD SHARING:
Plan to Share IPD: Yes
I will share all the documents related to the case.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: by2and half years
Access Criteria: the criteria will be discussed later